CLINICAL TRIAL: NCT03533192
Title: Teenage Pregnancy Prevention: Replication of Evidence-based Programs
Brief Title: Replication of Evidence-based Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: ETR Associates (Other); The Office of Adolescent Health, HHS (U.S. Federal Agency)
Responsible Party: Principal Investigator, Melissa Peskin, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSC-SPH-10-0455
Record Dates: First submitted 2018-04-23; First posted 2018-05-23 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Sexual Behavior
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data collectors were blind to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Receipt of It's Your Game...Keep it Real (Experimental): It's Your Game...Keep it Real is an HIV, STI, and teen pregnancy prevention program
  Interventions: Behavioral: It's Your Game...Keep it Real
- Usual care (No Intervention): Students received their regular health education.

INTERVENTIONS:
Behavioral: It's Your Game...Keep it Real — It's Your Game...Keep it Real consists of 12 50-minute lessons delivered in 7th grade (8 in class and 4 via computer) and 12 50-minute lessons delivered in 8th grade (7 in class and 5 via computer). In each grade, the curriculum integrates group-based classroom activities with personalized journaling and individually tailored computer-based activities. A life-skills decision-making paradigm (Select, Detect, Protect) underlies the activities, teaching students to select personal rules regarding risk behaviors, detect signs or situations that might challenge these rules, and use refusal skills and other tactics to protect these rules. The curriculum is grounded in social cognitive theory, the theory of triadic influence, and social influence models.
  Arms: Receipt of It's Your Game...Keep it Real

SUMMARY:
The purpose of this school-level randomized intervention trial is to evaluate the It's Your Game…Keep It Real program, an evidence-based teen pregnancy, HIV, and STI prevention program, among 2,000 students from 20 middle schools in 10 participating school districts in Harris County and surrounding areas. An audio computer-assisted self interview (A-CASI) assessment was used to assess demographic characteristics, psychosocial factors, sexual behaviors, and program exposure at three data collection points. Data was collected at baseline (preintervention), 6 months post intervention, and 12 months post intervention.

DETAILED DESCRIPTION:
Program Implemented: It's Your Game…Keep It Real (IYG) consists of 12 50-minute lessons delivered in 7th grade (8 in class and 4 via computer) and 12 50-minute lessons delivered in 8th grade (7 in class and 5 via computer). The intervention was provided to the same 7th and 8th graders over a two-year period (i.e., the same students receive up to 24 lessons over two years). The curriculum is grounded in social cognitive theory, the theory of triadic influence, and social influence models. The lessons were delivered according to the schedule that worked best for schools (for example, twice a week, once a week, or daily) within a school semester. The lessons were delivered by trained teachers during regular classroom time and were taught during a variety of subject areas (for example, physical education/health, social studies, and science). Teachers implementing the lessons were required to attend training in order to teach the 7th- and 8th-grade lessons.

Sample: This sample included students at 20 schools from selected school districts throughout the greater Houston, Texas, area that agreed to participate in the study and that served 7th and 8th grades. Student inclusion criteria required that students not face language barriers or require educational accommodations that would preclude them from participation in the survey data collection process. Data collection staff, blind to school study condition, recruited 7th-grade students attending eligible classes across the 20 middle schools participating in the randomized controlled trial. A mix of census and sampling was used when securing consent for participation. In schools with 250 or fewer 7th-grade students, consents were distributed to all students. For schools with 7th-grade enrollments of more than 250, classes were sampled randomly and consents were distributed to 180 students. The study included one cohort and followed students from 7th through 9th grades. The final enrolled sample size was 2,588 students for whom parental consent and student assent were obtained.

Setting: The study sites included 20 urban middle schools, in Harris County, Texas. The program was implemented in 10 intervention schools by trained facilitators. Most facilitators in both 7th and 8th grades were physical education teachers.

Data Collection: Data was collected at baseline (preintervention), 6 months post intervention, and 12 months post intervention.

Data Analysis: Impact data were analyzed using multilevel regression due to the nested nature of the study design (students within schools).

ELIGIBILITY:
Inclusion Criteria:

* enrolled in 7th grade at a participating school in fall 2012
* did not have limited capabilities or special needs as determined by the school
* spoke English well enough to understand the survey questions if they were read aloud.

Exclusion Criteria:

-did not meet inclusion criteria

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2588 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Initiation of vaginal or oral sex | 12 months after the program ends
  The variable is a yes/no measure of whether a person has ever had vaginal OR oral sex. The measure is created from the following items on the survey:
  * "Have you ever had sexual intercourse?" (defined in survey as penis in vagina)
  * "Have you ever had oral sex?" Participants who respond yes they have had sexual intercourse OR yes they have had oral sex are coded as 1 for yes; those who respond no they have not had sexual intercourse AND no they have not had oral sex are coded as 0 for no.

SECONDARY OUTCOMES:
Initiation of vaginal intercourse | 12 months after the program ends
  The variable is a yes/no measure of whether a person has ever had vaginal intercourse. The measure is based on the following item on the survey:
  • "Have you ever had sexual intercourse?" (defined in survey as penis in vagina) Respondents who respond yes they have had sexual intercourse are coded as 1 for yes and those who respond no they have not had vaginal intercourse are coded as 0 for no.
Initiation of oral sex | 12 months after the program ends
  The variable is a yes/no measure of whether a person has ever had oral sex. The measure is based on the following item on the survey:
  • "Have you ever had oral sex?" Respondents who respond yes they have had oral sex are coded as 1 for yes and those who respond no they have not had oral sex are coded as 0 for no.
Participation in vaginal sex without a condom | past 3 months
  The variable is a yes/no measure of whether a person participated in vaginal sex without a condom. It is only calculated for youth who reported having had sex in the past 3 months.
Participation in vaginal sex without an effective method of birth control | past 3 months
  The variable is a yes/no measure of whether a person participated in vaginal sex without an effective method of birth control. It is only calculated for youth who reported having had sex in the past 3 months.
Use of Condom at last sex | past 3 months
  The variable is a yes/no measure of whether a person reported using a condom the last time they had vaginal sex. It is only calculated for youth who reported having had sex in the past 3 months.
Use of effective method of birth control at last sex | past 3 months
  The variable is a yes/no measure of whether a person reported using an effective method of birth control the last time they had vaginal sex. It is only calculated for youth who reported having had sex in the past 3 months.
Percent of youth who report having vaginal sex 2 or more times in the past 3 months | past 3 months
  This variable is the percent of youth who reported having vaginal sex 2 or more times versus 1 time during the past 3 months. It is only calculated for youth who reported having had sex in the past 3 months.
Percent of youth who report having oral sex 2 or more times in the past 3 months | past 3 months
  This variable is the percent of youth who reported having oral sex 2 or more times versus 1 time during the past 3 months. It is only calculated for youth who reported having had sex in the past 3 months.
Percent of youth who report having vaginal sex with 2 or more partners in the past 3 months | past 3 months
  This variable is the percent of youth who reported having vaginal sex with 2 or more partners versus 1 partner during the last 3 months. It is only calculated for youth who reported having had sex in the past 3 months.
Percent of youth who report having oral sex with 2 or more partners in the past 3 months | past 3 months
  This variable is the percent of youth who reported having oral sex with 2 or more partners versus 1 partner during the last 3 months. It is only calculated for youth who reported having had sex in the past 3 months.
Percent of youth who report using drugs or alcohol before vaginal sex at least 1 time in the past 3 months | past 3 months
  This variable is the percent of youth who reported using drugs or alcohol before vaginal sex 1 time versus 0 times in the last 3 months. It is only calculated for youth who reported having had sex in the past 3 months.
Percent of youth who report using drugs or alcohol before oral sex at least 1 time in the past 3 months | past 3 months
  This variable is the percent of youth who reported using drugs or alcohol before oral sex 1 time versus 0 times in the last 3 months.It is only calculated for youth who reported having had sex in the past 3 months.
General condom knowledge | Past year
  This variable provides a mean score for general condom knowledge as measured by Coyle et al. (2014). Higher scores indicated greater condom knowledge. 6 items; yes, no, or not sure response format
General HIV/STI knowledge | Past year
  This variable provides a mean score for general HIV/STI knowledge as measured by Coyle et al. (1999). Higher scores indicated greater HIV/STI knowledge. 4 items; true, false, or not sure response format
Knowledge of signs and symptoms of STIs | Past year
  This variable provides a mean score for knowledge of signs and symptoms of STIs as measured by Coyle et al. (1999). Higher scores indicated greater knowledge of the signs and symptoms of STIs. 7 items; yes/no response format
General beliefs about waiting to have sex | Past year
  This variable provides a mean score for general beliefs about waiting to have sex as measured by Borawski et al. (2005). Higher scores reflect more positive beliefs about waiting to have sex; 4 items; 4-point scale (strongly disagree to strongly agree response format)
Beliefs about waiting until marriage to have sex | Past year
  This variable provides a mean score for beliefs about waiting until marriage to have sex as measured using items adapted from the Texas A&M High School Youth Survey and Teen Activities and Attitudes Survey; Higher scores reflect more positive beliefs about waiting until marriage to have sex; 3 items; 4-point scale (strongly disagree to strongly agree) response format
Reasons to not have sex | Past year
  This variable provides a mean score for the number of reasons participants provide for not having sex as measured by Coyle et al., 2004. A higher score reflects more reasons for not having sex. 10 items; Yes/No response format
General beliefs about condoms | Past year
  This variable provides a mean score for general beliefs about condoms as measured by the Case Western Health Promotion Study. A higher score reflects more positive beliefs about condoms. 3 items; 4-point scale (strongly disagree to strongly agree) response format
Perceived friends beliefs about waiting to have sex | Past year
  This variable provides a mean score for perceived friends beliefs about waiting to have sex as measured by Coyle et al., 2004. A higher score reflects students as being more likely to perceive their friends as having more negative attitudes towards waiting to have sex. 4 items; 4-point scale (strongly disagree to strongly agree) response format.
Perceived norms about sex (I) | Past year
  This variable provides a mean score that reflects a student's perception regarding how many teens who had sex wished they had waited until they were older (as measured by Coyle et al., 2004). A higher score means that a student perceived that more teens who had had sex wished they had waited until they were older; 1 item; 4-point scale (strongly disagree to strongly agree) response format
Perceived norms about sex (II) | Past year
  This variable provides a mean score that reflects a student's perception regarding how many other teens their age are having sex (as measured by Coyle et al., 2004). A higher score means that students perceived that many other teens their age were having sex; 1 item; 4-point scale (strongly disagree to strongly agree) response format
Perceived friends sexual behaviors (I) | Past year
  This variable provides a mean score that reflects a student's perception regarding how many of their friends have a boyfriend/girlfriend (as measured by Coyle et al., 2004). A higher score means that students perceived that many of their friends have a boyfriend/girlfriend; 1 item; 5-point scale (none to all) response format
Perceived friends sexual behaviors (II) | Past year
  This variable provides a mean score that reflects a student's perception regarding how many of their friends have had sex (as measured by Coyle et al., 2004). A higher score means that students perceived that many of their friends have had sex; 1 item; 5-point scale (none to all) response format
Perceived friends' beliefs about condoms | Past year
  This variable provides a mean score for perceived friends' beliefs about condoms as measured by the Case Western Health Promotion Study. A higher score reflects that students perceived their friends has having more positive beliefs about condoms. 3 items; 4-point scale (strongly disagree to strongly agree) response format
Perceived self-efficacy to refrain from having sex | Past year
  This variable provides a mean score for perceived self-efficacy to refrain from having sex (as measured by Coyle et al., 2004). A higher score reflects higher perceived self-efficacy to refrain from having sex. 6 items; 4 point scale (definitely could not to definitely could) response format
Perceived self-efficacy to negotiate the use of condoms with a partner | Past year
  This variable provides a mean score for perceived self-efficacy to negotiate the use of condoms with a partner as measured by Coyle et al., 2004. A higher score reflects greater self-efficacy. 2 items; 4-point scale (definitely could not to definitely could) response format
Perceived self-efficacy to obtain and correctly use condoms | Past year
  This variable provides a mean score for perceived self-efficacy to obtain and correctly use condoms as measured by Coyle et al., 2004. A higher score reflects greater self-efficacy. 3 items; 4-point scale (definitely could not to definitely could) response format
Personal limits regarding sex | Past year
  This variable provides a mean score for how one feels about how far he/she would go sexually and be able to communicate it to their partner as measured by Borawski et al., 2005. A higher score reflects that person would have higher perceived personal limits regarding sex. 1 item; 4-point scale (I have never really thought about how far I will go sexually to I know how far I would go sexually and I could tell a partner what I would do or not do)
Personal limits regarding condoms | Past year
  This variable provides a mean score for how one feels what he/she thinks about condom use and whether they could communicate it to a partner as measured by Borawski et al., 2005. A higher score reflects that person would have higher perceived personal limits regarding condoms. 1 item; 4-point scale (I have never really thought about using condoms to I know whether or not I would use condoms and I could tell my partner)
Communication with parents about sex | Past year
  This variable provides a mean score for parental communication about sex as measured by Ball et al., 2004 and Miller et al., 1998. A higher score reflects greater communication with parents. 6 items; 3-point scale (we've never talked about it to we've talked about it lots of times)
Exposure to risky situations | Past 3 months
  This variable provides a mean score for student exposure to risky situations as measured by Borawski et al., 2005 and Coyle et al., 2004. A higher score reflects more exposure to risky situations (e.g., gone to someone's house when an adult was not there). 5 items; 5-point scale (never to 6 times or more) response format
Intentions to have sex in the next year | Past year
  This variable provides a mean score for student intentions to have sex in the next year if they have the chance as measured by Tortolero et al., 2010. A higher score reflects greater intentions to have sex in the next year. 1 item; 4-point scale (yes, definitely to no, definitely not) response format
Intentions to remain abstinent until the end of high school | Past year
  This variable provides a mean score for student intentions remain abstinent until the end of high school as measured by the Case Western Health Promotion Study. A higher score reflects greater intentions to remain abstinent. 1 item; 4-point scale (yes, definitely to no, definitely not)
Intentions to remain abstinent until marriage | Past year
  This variable provides a mean score for student intentions to remain abstinent until marriage as measured by the Case Western Health Promotion Study. A higher score reflects greater intentions to remain abstinent until marriage. 1 item; 4-point scale (yes, definitely to no, definitely not)
Intentions to use a condom if have sex in the next year | Past year
  This variable provides a mean score for student intentions to use a condom if they have sex in the next year as measured by Tortolero et al., 2010. A higher score reflects greater intentions to use a condom; 1 item; 4-point scale (yes, definitely to no, definitely not)
Intentions to use effective birth control if have sex in the next year | Past year
  This variable provides a mean score for student intentions to use effective birth control if they have sex in the next year as measured by Tortolero et al., 2010. A higher score reflects greater intentions to use effective birth control; 1 item; 4-point scale (yes, definitely to no, definitely not)
Intentions to get tested for HIV/STI if think at risk | Past year
  This variable provides a mean score for student intentions to get tested for HIV/STI if they think they are at risk as measured by the Safer Choices survey. A higher score reflects greater intentions to get tested; 1 item; 4-point scale (yes, definitely to no, definitely not)

CONTACTS AND LOCATIONS:
Overall Officials: Susan T Emery, PhD, Principal Investigator — UT School of Public Health

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peskin MF, Coyle KK, Anderson PM, Laris BA, Glassman JR, Franks HM, Thiel MA, Potter SC, Unti T, Edwards S, Johnson-Baker K, Cuccaro PM, Diamond P, Markham CM, Shegog R, Baumler ER, Gabay EK, Emery ST. Replication of It's Your Game...Keep It Real! in Southeast Texas. J Prim Prev. 2019 Jun;40(3):297-323. doi: 10.1007/s10935-019-00549-0. PMID 31028508